CLINICAL TRIAL: NCT04800432
Title: ADAPT+: Optimizing an Intervention to Promote Healthy Behaviors in Rural, Latino Youth With Obesity and Their Parents, Using Mindfulness Strategies
Brief Title: Adapting Diet and Action for Everyone (ADAPT+)
Acronym: ADAPT+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00039979; R34AT010661 (NIH)
Record Dates: First submitted 2021-02-24; First posted 2021-03-16 (Actual); Results first posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Obesity
Keywords: Latino; Rural Communities; Mindfulness
MeSH Terms: conditions — Pediatric Obesity | interventions — Acclimatization

STUDY DESIGN:
Intervention Model Description: Aim 2 includes randomization to a comparison group - 48 parent-child dyads (96 individuals) anticipated for enrollment.
  Aim 2 was the small pilot RCT
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Feasibility and acceptability of ADAPT+ (Experimental): ADAPT+ is a family-based obesity intervention for high-risk Latino youth and their parents living in rural communities that incorporates culture-specific components and mindfulness-based approaches to promote adaptive health behaviors in a high-risk and underserved population.
  Interventions: Behavioral: ADAPT+
- Enhanced Usual Care (EUC) (Active Comparator): Enhanced Usual Care (EUC) provides publicly available material in both English and Spanish on the role of diet and exercise in pediatric obesity in a one-time information session.
  Interventions: Behavioral: EUC

INTERVENTIONS:
Behavioral: ADAPT+ — ADAPT+ is designed as an 6-week intervention. For each session, children and parents participate in separate 1.5-hour group meetings, followed by a joint goal setting session. Practical strategies related to improving diet and physical activity as well as the role of dealing with parent stress-related factors related to making long-lasting behavioral changes in the family are addressed.
  Arms: Feasibility and acceptability of ADAPT+
Behavioral: EUC — Enhanced Usual Care is an abbreviated version of the full ADAPT+ intervention in which parents are engaged in a one-time, two hour information session to also learn knowledge and skills to improve the health and lifestyle behaviors for their child and for themselves.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
The purpose of this study is to refine and optimize an obesity intervention with rural underserved Latino children and their parents that combines a standard family-based behavioral approach, the "gold standard" for pediatric obesity treatment, with a mindfulness approach focusing on stress reduction (now ADAPT+).

DETAILED DESCRIPTION:
Latino youth have the highest prevalence of obesity as compared to Black or White youth, and are at high risk for adult obesity-related complications including cardiovascular disease. Moreover, Latino youth living in rural communities have an increased risk of adult obesity and mortality due to obesity-related chronic disease than Latinos living elsewhere. The investigators synthesized the prior childhood obesity intervention and tailored the evidence informed, theory-based, multi-family behavioral intervention, Adapting Diet and Action for Everyone (ADAPT), to the acculturation status, language, and national origin of the target population - obese, school-aged (8-12 years old) Latino youth and their parents living in rural areas. However, because the role of parent stress on obesity has not been adequately addressed in interventions aimed at reducing obesity in Latino youth, it is argued that mindfulness parent stress reduction strategies may be a key component to improving eating and physical activity (PA) behaviors in both children and their parents. This study proposes a refinement and optimization of the original ADAPT obesity intervention protocol to include mindfulness parent stress reduction strategies (now ADAPT+) and feasibility assessment of ADAPT+ implementation.

Aim 1: Refinement of ADAPT+ (ADAPT + mindfulness parent stress reduction). Aim 1A and Aim 1B were focus groups with promotoras from the target communities and parents. The intervention manual was refined based on the qualitative feedback. Aim 1C further refines the manual via a small one parent-child cohort. Data collected at Aim 1C was used to finalize and optimize a culturally acceptable ADAPT+ evaluated in Aim 2.

Aim 2: Feasibility and Acceptability trial. A randomized trial testing feasibility of ADAPT+ vs. Enhanced Usual Care (EUC) conducted in two rural communities. It is anticipated that compared to EUC, ADAPT+ dyads will have a lower attrition rate and will report greater satisfaction. The investigators also explore whether the eating and stress indices are sensitive to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Child with a BMI %ile of 85 or higher.
* The target parent is at least 18 years old, is the main meal preparer, speaks and reads Spanish at a minimum of a 4th grade reading level (able to follow basic instructions in Spanish), and able to perform simple physical exercises.

Exclusion Criteria:

* A child who has a medical/developmental condition that precludes weight loss using conventional diet and PA methods.
* A child has been on antibiotics or steroids in the previous three months.
* The parent is ineligible if he/she is non-ambulatory, is pregnant, or has a medical condition that may be negatively impacted by PA.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2021-03-06 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Stern, PhD, Principal Investigator — University of South Florida
Locations (1):
- Hispanic Services Council, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of childhood and adult obesity in the United States, 2011-2012. JAMA. 2014 Feb 26;311(8):806-14. doi: 10.1001/jama.2014.732. PMID 24570244
- [Background] Lichter DT. Immigration and the New Racial Diversity in Rural America. Rural Sociol. 2012 Mar;77(1):3-35. doi: 10.1111/j.1549-0831.2012.00070.x. Epub 2012 Mar 1. PMID 26478602
- [Background] Bates LM, Acevedo-Garcia D, Alegria M, Krieger N. Immigration and generational trends in body mass index and obesity in the United States: results of the National Latino and Asian American Survey, 2002-2003. Am J Public Health. 2008 Jan;98(1):70-7. doi: 10.2105/AJPH.2006.102814. Epub 2007 Nov 29. PMID 18048787
- [Background] Haldeman GA, Croft JB, Giles WH, Rashidee A. Hospitalization of patients with heart failure: National Hospital Discharge Survey, 1985 to 1995. Am Heart J. 1999 Feb;137(2):352-60. doi: 10.1053/hj.1999.v137.95495. PMID 9924171
- [Background] Lutfiyya MN, Lipsky MS, Wisdom-Behounek J, Inpanbutr-Martinkus M. Is rural residency a risk factor for overweight and obesity for U.S. children? Obesity (Silver Spring). 2007 Sep;15(9):2348-56. doi: 10.1038/oby.2007.278. PMID 17890504
- [Background] Jilcott SB, Wade S, McGuirt JT, Wu Q, Lazorick S, Moore JB. The association between the food environment and weight status among eastern North Carolina youth. Public Health Nutr. 2011 Sep;14(9):1610-7. doi: 10.1017/S1368980011000668. Epub 2011 Apr 13. PMID 21486525
- [Background] Wang Y, Beydoun MA. The obesity epidemic in the United States--gender, age, socioeconomic, racial/ethnic, and geographic characteristics: a systematic review and meta-regression analysis. Epidemiol Rev. 2007;29:6-28. doi: 10.1093/epirev/mxm007. Epub 2007 May 17. PMID 17510091
- [Background] Butte NF, Cai G, Cole SA, Comuzzie AG. Viva la Familia Study: genetic and environmental contributions to childhood obesity and its comorbidities in the Hispanic population. Am J Clin Nutr. 2006 Sep;84(3):646-54; quiz 673-4. doi: 10.1093/ajcn/84.3.646. PMID 16960181
- [Background] Stovitz SD, Schwimmer JB, Martinez H, Story MT. Pediatric obesity: the unique issues in Latino-American male youth. Am J Prev Med. 2008 Feb;34(2):153-60. doi: 10.1016/j.amepre.2007.09.034. PMID 18201646
- [Background] Wenten M, Gilliland FD, Baumgartner K, Samet JM. Associations of weight, weight change, and body mass with breast cancer risk in Hispanic and non-Hispanic white women. Ann Epidemiol. 2002 Aug;12(6):435-4. doi: 10.1016/s1047-2797(01)00293-9. PMID 12160603
- [Background] Golan M, Crow S. Targeting parents exclusively in the treatment of childhood obesity: long-term results. Obes Res. 2004 Feb;12(2):357-61. doi: 10.1038/oby.2004.45. PMID 14981230
- [Background] Janicke DM, Steele RG, Gayes LA, Lim CS, Clifford LM, Schneider EM, Carmody JK, Westen S. Systematic review and meta-analysis of comprehensive behavioral family lifestyle interventions addressing pediatric obesity. J Pediatr Psychol. 2014 Sep;39(8):809-25. doi: 10.1093/jpepsy/jsu023. Epub 2014 May 13. PMID 24824614
- [Background] Isasi CR, Hua S, Jung M, Carnethon MR, Perreira K, Vidot DC, Salazar CR, McCurley JL, Sotres-Alvarez D, Van Horn L, Delamater AM, Llabre MM, Gallo LC. The Association of Parental/Caregiver Chronic Stress with Youth Obesity: Findings from the Study of Latino Youth and the Hispanic Community Health Study/Study of Latinos Sociocultural Ancillary Study. Child Obes. 2017 Aug;13(4):251-258. doi: 10.1089/chi.2016.0205. Epub 2017 Mar 1. PMID 28398853
- [Background] Tsenkova V, Boylan JM, Ryff C. Stress eating and health. Findings from MIDUS, a national study of US adults. Appetite. 2013 Oct;69:151-5. doi: 10.1016/j.appet.2013.05.020. Epub 2013 Jun 6. PMID 23747576
- [Background] Block JP, He Y, Zaslavsky AM, Ding L, Ayanian JZ. Psychosocial stress and change in weight among US adults. Am J Epidemiol. 2009 Jul 15;170(2):181-92. doi: 10.1093/aje/kwp104. Epub 2009 May 22. PMID 19465744
- [Background] Daly P, Pace T, Berg J, Menon U, Szalacha LA. A mindful eating intervention: A theory-guided randomized anti-obesity feasibility study with adolescent Latino females. Complement Ther Med. 2016 Oct;28:22-8. doi: 10.1016/j.ctim.2016.07.006. Epub 2016 Aug 1. PMID 27670866
- [Background] Dalen J, Brody JL, Staples JK, Sedillo D. A Conceptual Framework for the Expansion of Behavioral Interventions for Youth Obesity: A Family-Based Mindful Eating Approach. Child Obes. 2015 Oct;11(5):577-84. doi: 10.1089/chi.2014.0150. Epub 2015 Sep 1. PMID 26325143
- [Background] Onken LS, Carroll KM, Shoham V, Cuthbert BN, Riddle M. Reenvisioning Clinical Science: Unifying the Discipline to Improve the Public Health. Clin Psychol Sci. 2014 Jan 1;2(1):22-34. doi: 10.1177/2167702613497932. PMID 25821658
- [Background] Naar S, Czajkowski SM, Spring B. Innovative study designs and methods for optimizing and implementing behavioral interventions to improve health. Health Psychol. 2018 Dec;37(12):1081-1091. doi: 10.1037/hea0000657. Epub 2018 Oct 11. PMID 30307270
- [Background] Elder JP, Ayala GX, Parra-Medina D, Talavera GA. Health communication in the Latino community: issues and approaches. Annu Rev Public Health. 2009;30:227-51. doi: 10.1146/annurev.publhealth.031308.100300. PMID 19296776
- [Background] Ayala GX, Vaz L, Earp JA, Elder JP, Cherrington A. Outcome effectiveness of the lay health advisor model among Latinos in the United States: an examination by role. Health Educ Res. 2010 Oct;25(5):815-40. doi: 10.1093/her/cyq035. Epub 2010 Jul 5. PMID 20603384
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Pena MM, Dixon B, Taveras EM. Are you talking to ME? The importance of ethnicity and culture in childhood obesity prevention and management. Child Obes. 2012 Feb;8(1):23-7. doi: 10.1089/chi.2011.0109. PMID 22799474
- [Background] Singh GK, Siahpush M, Kogan MD. Rising social inequalities in US childhood obesity, 2003-2007. Ann Epidemiol. 2010 Jan;20(1):40-52. doi: 10.1016/j.annepidem.2009.09.008. PMID 20006275
- [Background] Biener AI, Cawley J, Meyerhoefer C. The medical care costs of obesity and severe obesity in youth: An instrumental variables approach. Health Econ. 2020 May;29(5):624-639. doi: 10.1002/hec.4007. Epub 2020 Feb 23. PMID 32090412
- [Background] Warne JP. Shaping the stress response: interplay of palatable food choices, glucocorticoids, insulin and abdominal obesity. Mol Cell Endocrinol. 2009 Mar 5;300(1-2):137-46. doi: 10.1016/j.mce.2008.09.036. Epub 2008 Oct 15. PMID 18984030
- [Background] van Jaarsveld CH, Fidler JA, Steptoe A, Boniface D, Wardle J. Perceived stress and weight gain in adolescence: a longitudinal analysis. Obesity (Silver Spring). 2009 Dec;17(12):2155-61. doi: 10.1038/oby.2009.183. Epub 2009 Jun 11. PMID 19521353
- [Background] Lissau I, Sorensen TI. Parental neglect during childhood and increased risk of obesity in young adulthood. Lancet. 1994 Feb 5;343(8893):324-7. doi: 10.1016/s0140-6736(94)91163-0. PMID 7905145
- [Background] Hughes SO, Power TG, Liu Y, Sharp C, Nicklas TA. Parent emotional distress and feeding styles in low-income families. The role of parent depression and parenting stress. Appetite. 2015 Sep;92:337-42. doi: 10.1016/j.appet.2015.06.002. Epub 2015 Jun 4. PMID 26050915
- [Background] Urizar GG, Hurtz SQ, Ahn DK, King AC, Albright CL, Atienza AA. Influence of maternal stress on successful participation in a physical activity intervention: the IMPACT Project. Women Health. 2005;42(4):63-82. doi: 10.1300/j013v42n04_04. PMID 16782676
- [Background] Dallman MF, Pecoraro N, Akana SF, La Fleur SE, Gomez F, Houshyar H, Bell ME, Bhatnagar S, Laugero KD, Manalo S. Chronic stress and obesity: a new view of "comfort food". Proc Natl Acad Sci U S A. 2003 Sep 30;100(20):11696-701. doi: 10.1073/pnas.1934666100. Epub 2003 Sep 15. PMID 12975524
- [Background] Romero AJ. A pilot test of the Latin active hip hop intervention to increase physical activity among low-income Mexican-American adolescents. Am J Health Promot. 2012 Mar-Apr;26(4):208-11. doi: 10.4278/ajhp.090123-ARB-24. PMID 22375569
- [Background] Olvera N, Bush JA, Sharma SV, Knox BB, Scherer RL, Butte NF. BOUNCE: a community-based mother-daughter healthy lifestyle intervention for low-income Latino families. Obesity (Silver Spring). 2010 Feb;18 Suppl 1:S102-4. doi: 10.1038/oby.2009.439. PMID 20107454
- [Background] Barkin SL, Gesell SB, Poe EK, Ip EH. Changing overweight Latino preadolescent body mass index: the effect of the parent-child dyad. Clin Pediatr (Phila). 2011 Jan;50(1):29-36. doi: 10.1177/0009922810379039. Epub 2010 Sep 13. PMID 20837625
- [Background] Summerbell CD, Waters E, Edmunds LD, Kelly S, Brown T, Campbell KJ. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD001871. doi: 10.1002/14651858.CD001871.pub2. PMID 16034868
- [Background] Skelton JA, Buehler C, Irby MB, Grzywacz JG. Where are family theories in family-based obesity treatment?: conceptualizing the study of families in pediatric weight management. Int J Obes (Lond). 2012 Jul;36(7):891-900. doi: 10.1038/ijo.2012.56. Epub 2012 Apr 24. PMID 22531090
- [Background] Sosa ET. Mexican American mothers' perceptions of childhood obesity: a theory-guided systematic literature review. Health Educ Behav. 2012 Aug;39(4):396-404. doi: 10.1177/1090198111398129. Epub 2011 May 6. PMID 21551423
- [Background] Allen ML, Elliott MN, Morales LS, Diamant AL, Hambarsoomian K, Schuster MA. Adolescent participation in preventive health behaviors, physical activity, and nutrition: differences across immigrant generations for Asians and Latinos compared with Whites. Am J Public Health. 2007 Feb;97(2):337-43. doi: 10.2105/AJPH.2005.076810. Epub 2006 Nov 30. PMID 17138919
- [Background] Sussner KM, Lindsay AC, Greaney ML, Peterson KE. The influence of immigrant status and acculturation on the development of overweight in Latino families: a qualitative study. J Immigr Minor Health. 2008 Dec;10(6):497-505. doi: 10.1007/s10903-008-9137-3. PMID 18373200
- [Background] Popkin BM, Udry JR. Adolescent obesity increases significantly in second and third generation U.S. immigrants: the National Longitudinal Study of Adolescent Health. J Nutr. 1998 Apr;128(4):701-6. doi: 10.1093/jn/128.4.701. PMID 9521631
- [Background] Martinez SM, Rhee K, Blanco E, Boutelle K. Maternal attitudes and behaviors regarding feeding practices in elementary school-aged Latino children: a pilot qualitative study on the impact of the cultural role of mothers in the US-Mexican border region of San Diego, California. J Acad Nutr Diet. 2014 Feb;114(2):230-237. doi: 10.1016/j.jand.2013.09.028. Epub 2013 Dec 4. PMID 24315129
- [Background] Baughcum AE, Burklow KA, Deeks CM, Powers SW, Whitaker RC. Maternal feeding practices and childhood obesity: a focus group study of low-income mothers. Arch Pediatr Adolesc Med. 1998 Oct;152(10):1010-4. doi: 10.1001/archpedi.152.10.1010. PMID 9790612
- [Background] Reifsnider E, Flores-Vela AR, Beckman-Mendez D, Nguyen H, Keller C, Dowdall-Smith S. Perceptions of children's body sizes among mothers living on the Texas-Mexico border (La Frontera). Public Health Nurs. 2006 Nov-Dec;23(6):488-95. doi: 10.1111/j.1525-1446.2006.00588.x. PMID 17096773
- [Background] Shonkoff ET, Dunton GF, Chou CP, Leventhal AM, Bluthenthal R, Pentz MA. Direct and indirect effects of parent stress on child obesity risk and added sugar intake in a sample of Southern California adolescents. Public Health Nutr. 2017 Dec;20(18):3285-3294. doi: 10.1017/S136898001700252X. Epub 2017 Oct 5. PMID 28980520
- [Background] Nyklicek I, Mommersteeg PM, Van Beugen S, Ramakers C, Van Boxtel GJ. Mindfulness-based stress reduction and physiological activity during acute stress: a randomized controlled trial. Health Psychol. 2013 Oct;32(10):1110-3. doi: 10.1037/a0032200. Epub 2013 Mar 25. PMID 23527521
- [Background] Coatsworth JD, Duncan LG, Nix RL, Greenberg MT, Gayles JG, Bamberger KT, Berrena E, Demi MA. Integrating mindfulness with parent training: effects of the Mindfulness-Enhanced Strengthening Families Program. Dev Psychol. 2015 Jan;51(1):26-35. doi: 10.1037/a0038212. Epub 2014 Nov 3. PMID 25365122
- [Background] Olson KL, Emery CF. Mindfulness and weight loss: a systematic review. Psychosom Med. 2015 Jan;77(1):59-67. doi: 10.1097/PSY.0000000000000127. PMID 25490697
- [Background] Rogers JM, Ferrari M, Mosely K, Lang CP, Brennan L. Mindfulness-based interventions for adults who are overweight or obese: a meta-analysis of physical and psychological health outcomes. Obes Rev. 2017 Jan;18(1):51-67. doi: 10.1111/obr.12461. Epub 2016 Nov 11. PMID 27862826
- [Background] Kristeller JL, Wolever RQ. Mindfulness-based eating awareness training for treating binge eating disorder: the conceptual foundation. Eat Disord. 2011 Jan-Feb;19(1):49-61. doi: 10.1080/10640266.2011.533605. PMID 21181579
- [Background] Dumas JE. Mindfulness-based parent training: strategies to lessen the grip of automaticity in families with disruptive children. J Clin Child Adolesc Psychol. 2005 Dec;34(4):779-91. doi: 10.1207/s15374424jccp3404_20. PMID 16232075
- [Background] Halperin DT, Laux J, LeFranc-Garcia C, Araujo C, Palacios C. Findings From a Randomized Trial of Weight Gain Prevention Among Overweight Puerto Rican Young Adults. J Nutr Educ Behav. 2019 Feb;51(2):205-216. doi: 10.1016/j.jneb.2018.07.014. Epub 2018 Oct 2. PMID 30291016
- [Background] Coatsworth JD, Duncan LG, Greenberg MT, Nix RL. Changing Parent's Mindfulness, Child Management Skills and Relationship Quality With Their Youth: Results From a Randomized Pilot Intervention Trial. J Child Fam Stud. 2010 Apr 1;19(2):203-217. doi: 10.1007/s10826-009-9304-8. PMID 24013587
- [Background] Duncan LG, Coatsworth JD, Greenberg MT. A model of mindful parenting: implications for parent-child relationships and prevention research. Clin Child Fam Psychol Rev. 2009 Sep;12(3):255-70. doi: 10.1007/s10567-009-0046-3. PMID 19412664
- [Background] Jastreboff AM, Chaplin TM, Finnie S, Savoye M, Stults-Kolehmainen M, Silverman WK, Sinha R. Preventing Childhood Obesity Through a Mindfulness-Based Parent Stress Intervention: A Randomized Pilot Study. J Pediatr. 2018 Nov;202:136-142.e1. doi: 10.1016/j.jpeds.2018.07.011. Epub 2018 Sep 18. PMID 30241766
- [Background] Dahmer S. Do you have any advice on how to help with this problem of access to CAM therapies for patients without financial resources? Explore (NY). 2007 Sep-Oct;3(5):546. doi: 10.1016/j.explore.2007.07.013. No abstract available. PMID 17905369
- [Background] Stern M, Ewing L, Davila E, Thompson AL, Hale G, Mazzeo S. Design and rationale for NOURISH-T: a randomized control trial targeting parents of overweight children off cancer treatment. Contemp Clin Trials. 2015 Mar;41:227-37. doi: 10.1016/j.cct.2014.12.018. Epub 2015 Jan 2. PMID 25559916
- [Background] Mazzeo SE, Kelly NR, Stern M, Gow RW, Serdar K, Evans RK, Jones RM, Bulik CM. Nourishing Our Understanding of Role Modeling to Improve Support and Health (NOURISH): design and methods. Contemp Clin Trials. 2012 May;33(3):515-22. doi: 10.1016/j.cct.2012.01.003. Epub 2012 Jan 18. PMID 22273843
- [Background] Mazzeo SE, Kelly NR, Stern M, Gow RW, Cotter EW, Thornton LM, Evans RK, Bulik CM. Parent skills training to enhance weight loss in overweight children: evaluation of NOURISH. Eat Behav. 2014 Apr;15(2):225-9. doi: 10.1016/j.eatbeh.2014.01.010. Epub 2014 Feb 3. PMID 24854808
- [Background] Whitlock EP, O'Connor EA, Williams SB, Beil TL, Lutz KW. Effectiveness of weight management interventions in children: a targeted systematic review for the USPSTF. Pediatrics. 2010 Feb;125(2):e396-418. doi: 10.1542/peds.2009-1955. Epub 2010 Jan 18. PMID 20083531
- [Background] Skelton JA, Beech BM. Attrition in paediatric weight management: a review of the literature and new directions. Obes Rev. 2011 May;12(5):e273-81. doi: 10.1111/j.1467-789X.2010.00803.x. Epub 2010 Sep 29. PMID 20880126
- [Background] Perez LG, Arredondo EM, Elder JP, Barquera S, Nagle B, Holub CK. Evidence-based obesity treatment interventions for Latino adults in the U.S.: a systematic review. Am J Prev Med. 2013 May;44(5):550-60. doi: 10.1016/j.amepre.2013.01.016. PMID 23597822
- [Background] Bean MK, Wilson DB, Thornton LM, Kelly N, Mazzeo SE. Dietary intake in a randomized-controlled pilot of NOURISH: a parent intervention for overweight children. Prev Med. 2012 Sep;55(3):224-7. doi: 10.1016/j.ypmed.2012.06.016. Epub 2012 Jun 24. PMID 22735041
- [Background] Stern M, Bleck J, Ewing LJ, Davila E, Lynn C, Hale G, Mazzeo S. NOURISH-T: Targeting caregivers to improve health behaviors in pediatric cancer survivors with obesity. Pediatr Blood Cancer. 2018 May;65(5):e26941. doi: 10.1002/pbc.26941. Epub 2018 Jan 19. PMID 29350459
- [Background] Steiner-Adair C, Sjostrom L, Franko DL, Pai S, Tucker R, Becker AE, Herzog DB. Primary prevention of risk factors for eating disorders in adolescent girls: learning from practice. Int J Eat Disord. 2002 Dec;32(4):401-11. doi: 10.1002/eat.10089. PMID 12386905
- [Background] Austin SB. Prevention research in eating disorders: theory and new directions. Psychol Med. 2000 Nov;30(6):1249-62. doi: 10.1017/s0033291799002573. PMID 11097066
- [Background] Taylor SJ, Whincup PH, Hindmarsh PC, Lampe F, Odoki K, Cook DG. Performance of a new pubertal self-assessment questionnaire: a preliminary study. Paediatr Perinat Epidemiol. 2001 Jan;15(1):88-94. doi: 10.1046/j.1365-3016.2001.00317.x. PMID 11237120
- [Background] Galanti GA. The Hispanic family and male-female relationships: an overview. J Transcult Nurs. 2003 Jul;14(3):180-5. doi: 10.1177/1043659603014003004. PMID 12861920
- [Background] Wang JB, Cadmus-Bertram LA, Natarajan L, White MM, Madanat H, Nichols JF, Ayala GX, Pierce JP. Wearable Sensor/Device (Fitbit One) and SMS Text-Messaging Prompts to Increase Physical Activity in Overweight and Obese Adults: A Randomized Controlled Trial. Telemed J E Health. 2015 Oct;21(10):782-92. doi: 10.1089/tmj.2014.0176. Epub 2015 Jun 2. PMID 26431257
- [Background] Flynn MA, McNeil DA, Maloff B, Mutasingwa D, Wu M, Ford C, Tough SC. Reducing obesity and related chronic disease risk in children and youth: a synthesis of evidence with 'best practice' recommendations. Obes Rev. 2006 Feb;7 Suppl 1:7-66. doi: 10.1111/j.1467-789X.2006.00242.x. PMID 16371076
- [Background] Campbell M, Fitzpatrick R, Haines A, Kinmonth AL, Sandercock P, Spiegelhalter D, Tyrer P. Framework for design and evaluation of complex interventions to improve health. BMJ. 2000 Sep 16;321(7262):694-6. doi: 10.1136/bmj.321.7262.694. No abstract available. PMID 10987780
- [Background] Castro FG, Barrera M Jr, Martinez CR Jr. The cultural adaptation of prevention interventions: resolving tensions between fidelity and fit. Prev Sci. 2004 Mar;5(1):41-5. doi: 10.1023/b:prev.0000013980.12412.cd. PMID 15058911
- [Background] Palmberg AA, Stern M, Kelly NR, Bulik C, Belgrave FZ, Trapp SK, Hofmeier SM, Mazzeo SE. Adolescent Girls and Their Mothers Talk About Experiences of Binge and Loss of Control Eating. J Child Fam Stud. 2014 Nov;23(8):1403-1416. doi: 10.1007/s10826-013-9797-z. PMID 25400491
- [Background] Stunkard AJ, Sorensen T, Schulsinger F. Use of the Danish Adoption Register for the study of obesity and thinness. Res Publ Assoc Res Nerv Ment Dis. 1983;60:115-20. No abstract available. PMID 6823524
- [Background] Hendrickson KL, Rasmussen EB. Mindful eating reduces impulsive food choice in adolescents and adults. Health Psychol. 2017 Mar;36(3):226-235. doi: 10.1037/hea0000440. Epub 2016 Nov 3. PMID 27808529
- [Background] Levoy E, Lazaridou A, Brewer J, Fulwiler C. An exploratory study of Mindfulness Based Stress Reduction for emotional eating. Appetite. 2017 Feb 1;109:124-130. doi: 10.1016/j.appet.2016.11.029. Epub 2016 Nov 24. PMID 27890474
- [Background] Redwine LS, Henry BL, Pung MA, Wilson K, Chinh K, Knight B, Jain S, Rutledge T, Greenberg B, Maisel A, Mills PJ. Pilot Randomized Study of a Gratitude Journaling Intervention on Heart Rate Variability and Inflammatory Biomarkers in Patients With Stage B Heart Failure. Psychosom Med. 2016 Jul-Aug;78(6):667-76. doi: 10.1097/PSY.0000000000000316. PMID 27187845
- [Background] Redwine LS, Tsuang M, Rusiewicz A, Pandzic I, Cammarata S, Rutledge T, Hong S, Linke S, Mills PJ. A pilot study exploring the effects of a 12-week t'ai chi intervention on somatic symptoms of depression in patients with heart failure. J Altern Complement Med. 2012 Aug;18(8):744-8. doi: 10.1089/acm.2011.0314. Epub 2012 Jul 30. PMID 22845485
- [Background] Linke SE, Noble M, Hurst S, Strong DR, Redwine L, Norman SB, Lindamer LA. An Exercise-Based Program for Veterans with Substance Use Disorders: Formative Research. J Psychoactive Drugs. 2015 Jul-Aug;47(3):248-57. doi: 10.1080/02791072.2015.1047915. Epub 2015 Jun 22. PMID 26098629
- [Background] Wilson KL, Tomfohr L, Edwards K, Knott C, Hong S, Redwine L, Calfas K, Rock CL, von Kanel R, Mills PJ. Effects of Aerobic Fitness and Adiposity on Coagulation Biomarkers in Men vs. Women with Elevated Blood Pressure. Eur J Cardiovasc Med. 2012 Sep;2(2):122-128. Epub 2012 Sep 24. PMID 23105963
- [Background] Ammerman A, Leung MM, Cavallo D. Addressing disparities in the obesity epidemic. N C Med J. 2006 Jul-Aug;67(4):301-4. No abstract available. PMID 17066662
- [Background] Stewart DA, Carter JC, Drinkwater J, Hainsworth J, Fairburn CG. Modification of eating attitudes and behavior in adolescent girls: A controlled study. Int J Eat Disord. 2001 Mar;29(2):107-18. doi: 10.1002/1098-108x(200103)29:23.0.co;2-1. PMID 11429973
- [Background] Bracero W. Intimidades: confianza, gender, and hierarchy in the construction of Latino-Latina therapeutic relationships. Cult Divers Ment Health. 1998;4(4):264-77. PMID 9818515
- [Background] Lescano CM, Brown LK, Raffaelli M, Lima LA. Cultural factors and family-based HIV prevention intervention for Latino youth. J Pediatr Psychol. 2009 Nov-Dec;34(10):1041-52. doi: 10.1093/jpepsy/jsn146. Epub 2009 Jan 30. PMID 19181820
- [Background] Koskan A, Friedman DB, Messias DK, Brandt HM, Walsemann K. Sustainability of promotora initiatives: program planners' perspectives. J Public Health Manag Pract. 2013 Sep-Oct;19(5):E1-9. doi: 10.1097/PHH.0b013e318280012a. PMID 23295409
- [Background] London L, Hurtado-de-Mendoza A, Song M, Nagirimadugu A, Luta G, Sheppard VB. Motivators and barriers to Latinas' participation in clinical trials: the role of contextual factors. Contemp Clin Trials. 2015 Jan;40:74-80. doi: 10.1016/j.cct.2014.11.013. Epub 2014 Nov 26. PMID 25433203
- [Background] Leung, MM, Cavalcanti, OB, El Dada, A, Brown, M, Mateo, MF, Yeh MC. Treating Obesity in Latino Children: A Systematic Review of Current Interventions. International Journal of Child Health and Nutrition. 2017;6(1):1-15.
- [Background] Stern M, Lescano, C., Lopez Castillo, H., Lynn, C., & Bleck, J. Adaptando Dieta y Accion Para Todos (ADAPT): Targeting diet and physical activity of Latinos living in rural communities in Florida. In I. B. Thurston (chair). Culturally Responsive Assessments and Interventions to Address Pediatric Obesity: A Collaborative Symposium of the Diversity and Obesity SIGs. Society of Pediatric Psychology; 2017; Portland, OR.
- [Background] Stern M, Soca Lozano S, Lescano C, Rodriguez C, Redwine L. Developing Adaptando Dieta Y Accion Para Todos (ADAPT): An Intervention to Improve Healthy Lifestyle Behaviors Among Latino Parents and Children Living in Rural Communities. J Immigr Minor Health. 2021 Feb;23(1):88-94. doi: 10.1007/s10903-020-01037-y. PMID 32533505
- [Background] Black DS, Fernando R. Mindfulness Training and Classroom Behavior Among Lower-Income and Ethnic Minority Elementary School Children. J Child Fam Stud. 2014 Oct;23(7):1242-1246. doi: 10.1007/s10826-013-9784-4. PMID 25624749
- [Background] U. S. Census Bureau. American Community Survey. Author. https://www.census.gov/programs-surveys/acs/data.html. Published 2013.
- [Background] Bolin JN, Bellamy G, Ferdinand AO, Kash BA, Helduser JW. Rural Healthy People 2020. Vol 1. College Station, TX: Texas A&M Health Science Center School of Public Health, Southwest Rural Health Research Center. http://sph.tamhsc.edu/srhrc/docs/rhp2020-volume-1.pdf; 2015.
- [Background] Gutman, L. M., McLoyd, V. C., & Tokoyawa, T. (2005). Financial strain, neighborhood stress, parenting behaviors, and adolescent adjustment in urban African American families. Journal of Research on Adolescence, 15(4), 425-449. https://doi.org/10.1111/j.1532-7795.2005.00106.x
- [Background] Haldeman LA, Gruber KJ, Ingram KP. Determinants of food security and diet among rural and urban Latino/Hispanic immigrants. J Hunger Environ Nutr. 2008;2(4):67-83.
- [Background] Del Parigi A. Neuroanatomical correlates of hunger and satiety in lean and obese individuals. In: Dube L, Bechara A, Dagher A, et al., eds. Obesity Prevention. Academic Press; 2010:253-271.
- [Background] Kabat-Zinn J. Mindfulness-based interventions in context: past, present, and future. Clinical psychology: Science and practice. 2003;10(2):144-156.
- [Derived] Stern M, Rancourt D, Soca Lozano S, Buro AW, Gray HL, Rodriguez C, Bailey R, Redwine L. Delivering ADAPT+ to Latino Families Living in Rural Communities: Feasibility and Acceptability of Implementing a Health Promotion Program Including Mindfulness. J Pediatr Psychol. 2023 Aug 29;48(8):666-675. doi: 10.1093/jpepsy/jsad049. PMID 37541829

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 48 parent/child dyad pairs were considered enrolled in the study.
Groups:
- Feasibility and Acceptability of ADAPT+: ADAPT+ is a family-based obesity intervention for high-risk Latino youth and their parents living in rural communities that incorporates culture-specific components and mindfulness-based approaches to promote adaptive health behaviors in a high-risk and underserved population.
  ADAPT+: ADAPT+ is designed as a 6-week intervention. For each session, children and parents participate in separate 1.5-hour group meetings, followed by a joint goal-setting session. Practical strategies related to improving diet and physical activity as well as the role of dealing with parent stress-related factors related to making long-lasting behavioral changes in the family are addressed.
Period: Overall Study
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Started | 47 | 48
Parents Who Started | 24 | 24
Youth Who Started | 23 (One parent attended baseline without the youth.) | 24
Completed | 41 | 35
Not Completed | 6 | 13

BASELINE CHARACTERISTICS:
Groups:
- Feasibility and Acceptability of ADAPT+: ADAPT+ is a family-based obesity intervention for high-risk Latino youth and their parents living in rural communities that incorporates culture-specific components and mindfulness-based approaches to promote adaptive health behaviors in a high-risk and underserved population.
  ADAPT+: ADAPT+ is designed as an 8-week intervention. For each session, children and parents participate in separate 1.5-hour group meetings, followed by a joint goal setting session. Practical strategies related to improving diet and physical activity as well as the role of dealing with parent stress-related factors related to making long-lasting behavioral changes in the family are addressed.
- Total: Total of all reporting groups
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 47 | 48 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall number of participants includes both parents and children participating in the study. A row was created for each group (i.e., one row for parents and one row for children), in order to report Mean and SD values accordingly.
  years
    Parents: number analyzed (Participants) | 24 | 24 | 48
    Parents | 39.60 (7.19) | 38.56 (6.92) | 38.98 (7.01)
    Youth: number analyzed (Participants) | 23 | 24 | 47
    Youth | 9.61 (1.55) | 10.36 (1.45) | 9.99 (1.53)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The overall number of participants represents participating parents and children. Row population was created to represent each age group (e.g., parents, youth).
  Participants
    Parents: number analyzed (Participants) | 24 | 24 | 48
    Parents: Female | 23 | 21 | 44
    Parents: Male | 1 | 3 | 4
    Youth: number analyzed (Participants) | 23 | 24 | 47
    Youth: Female | 11 | 13 | 24
    Youth: Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 47 | 48 | 95
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The overall number of participants represents participating parents and children. Row population was created to represent each age group (e.g., parents, youth).
  Participants
    Parents: number analyzed (Participants) | 24 | 24 | 48
    Parents: White | 16 | 14 | 30
    Parents: Black | 0 | 1 | 1
    Parents: More than one race | 5 | 3 | 8
    Parents: Other race | 1 | 4 | 5
    Parents: Unknown | 2 | 2 | 4
    Youth: number analyzed (Participants) | 23 | 24 | 47
    Youth: White | 16 | 13 | 29
    Youth: Black | 0 | 1 | 1
    Youth: More than one race | 5 | 3 | 8
    Youth: Other race | 1 | 4 | 5
    Youth: Unknown | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 95
BMI (parent) [Mean (Standard Deviation); unit: kg/m^2] — Population: Row population differs from Overall because BMI was only calculated for participating parents.
  kg/m^2
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 31.68 (4.88) | 31.18 (5.68) | 31.43 (5.25)
BMI z-score (child) [Mean (Standard Deviation); unit: Z-score] — Z Body Mass Index (BMI). 0 represents the population mean. The higher the score, the higher the BMI, based on age and gender. There are no established clinically relevant thresholds for z-BMI. Population: Row population differs from Overall because z-BMI was only calculated for participating children.
  Z-score
    number analyzed (Participants) | 24 | 18 | 42
    (all) | 2.25 (.91) | 1.69 (1.05) | 1.96 (1.01)
Waist-to-hip ratio (WHR) (parent) [Mean (Standard Deviation); unit: Waist-to-hip ratio] — Population: Row population differs from Overall because this variable represents the waist-to-hip ratio for participating parents only.
  Waist-to-hip ratio
    number analyzed (Participants) | 24 | 24 | 48
    (all) | .90 (.05) | .90 (.07) | .90 (.06)
Waist-to-hip ratio (WHR) (child) [Mean (Standard Deviation); unit: Waist-to-hip ratio] — Population: Row population differs from Overall because this variable represents the waist-to-hip ratio for participating children only.
  Waist-to-hip ratio
    number analyzed (Participants) | 24 | 18 | 42
    (all) | .92 (.06) | .90 (.08) | .91 (.07)
Resting blood pressure (parent) [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Population: Row population differs from Overall because this variable represents the blood pressure data for participating parents only.
  millimeters of mercury (mmHg)
    Systolic Blood Pressure: number analyzed (Participants) | 24 | 24 | 48
    Systolic Blood Pressure | 119.40 (15.27) | 117.17 (15.45) | 118.28 (15.24)
    Diastolic Blood Pressure: number analyzed (Participants) | 24 | 24 | 48
    Diastolic Blood Pressure | 72.39 (8.87) | 71.21 (9.94) | 71.80 (9.34)
Resting blood pressure (child) [Mean (Standard Deviation); unit: millimeters of mercury (mmHg)] — Population: Row population differs from Overall because this variable represents the blood pressure data for participating children only.
  millimeters of mercury (mmHg)
    Systolic Blood Pressure: number analyzed (Participants) | 23 | 24 | 47
    Systolic Blood Pressure | 108.34 (9.50) | 105.67 (10.60) | 106.96 (10.05)
    Diastolic Blood Pressure: number analyzed (Participants) | 23 | 24 | 47
    Diastolic Blood Pressure | 61.00 (6.61) | 57.92 (9.23) | 59.43 (8.12)
Child Sugar Sweet Beverage and Fast Food Intake Instrument (child) [Mean (Standard Deviation); unit: units on a scale] — 11 items on food and physical activity behaviors for youth. Fruit & Veg Frequency: 0-15, higher scores mean fruits and veggies consumed more frequently.
  Fruit & Veg Quantity: 0-5, higher scores mean larger fruit and veggie quantity consumed.
  Sugar-Sweetened Beverage Freq (SSB): 0-8, higher scores mean SSB consumed more frequently.
  Sugar-Sweetened Beverage Quantity: 0-5, higher scores mean larger quantities of SSB consumed.
  Fast Food Frequency: 0-4, higher scores mean fast food consumed more frequently.
  Fast Food Quantity: 0-16, higher scores mean larger quantities of fast food consumed. Population: Row population differs from Overall because this measure was only assessed in participating children.
  units on a scale
    Sugar-Sweetened Beverage: Frequency: number analyzed (Participants) | 23 | 24 | 47
    Sugar-Sweetened Beverage: Frequency | 2.37 (2.16) | 2.39 (1.61) | 2.38 (1.86)
    Sugar-Sweetened Beverage: Quantity: number analyzed (Participants) | 23 | 24 | 47
    Sugar-Sweetened Beverage: Quantity | 2.06 (1.26) | 1.96 (.80) | 2.00 (1.03)
    Fast Food: Frequency: number analyzed (Participants) | 23 | 24 | 47
    Fast Food: Frequency | 1.00 (.76) | .78 (.54) | .88 (.65)
    Fast Food: Quantity: number analyzed (Participants) | 23 | 24 | 47
    Fast Food: Quantity | 3.81 (2.07) | 3.17 (2.68) | 3.47 (2.40)
    Fruit & Vegetable: Frequency: number analyzed (Participants) | 23 | 24 | 47
    Fruit & Vegetable: Frequency | 7.31 (3.18) | 6.44 (3.63) | 6.85 (3.40)
    Fruit & Vegetable: Quantity: number analyzed (Participants) | 23 | 24 | 47
    Fruit & Vegetable: Quantity | 3.34 (.72) | 3.25 (.79) | 3.29 (.75)
Stephenson Multigroup Acculturation Scale [SMAS] (parent) [Mean (Standard Deviation); unit: units on a scale] — Population: Row population differs from Overall because this variable represents the acculturation data asked only to participating parents.
  units on a scale
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 3.00 (.36) | 2.99 (.37) | 2.99 (.36)
Latino Dietary Behaviors Questionnaire (parent) [Mean (Standard Deviation); unit: units on a scale] — Population: Row population differs from Overall because this measure was only assessed in participating parents.
  units on a scale
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 24.96 (4.65) | 24.83 (4.00) | 24.90 (4.29)
Perceived Stress Scale (PSS) (parent) [Mean (Standard Deviation); unit: units on a scale] — Population: Row population differs from Overall because this measure was only assessed in participating parents.
  units on a scale
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 18.13 (5.78) | 16.04 (6.79) | 17.08 (6.32)
Recognize subscale of the Mindful Eating Questionnaire (parent) [Mean (Standard Deviation); unit: units on a scale] — Population: Row population differs from Overall because this measure was only assessed in participating parents.
  units on a scale
    number analyzed (Participants) | 24 | 24 | 48
    (all) | 29.79 (4.35) | 29.83 (3.67) | 29.81 (3.98)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Acceptability was measured by a program satisfaction survey at the end of the intervention. Items were rated on a scale from 1 (Not at all) to 4 (Very) enjoyable, comfortable, receptive, relevant, or helpful, depending on the item's content. A mean score was calculated using all items to reflect overall satisfaction, with higher scores indicating greater satisfaction. Only parents completed the program satisfaction survey.
  Minimum score: 1 Maximum score: 4 Higher scores mean better outcomes.
Time Frame: 6 weeks after baseline
Population: This number refers to the parents who completed the exit survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 18
score on a scale | 3.91 (.18) | 3.85 (.32)

2. Primary Outcome: Feasibility - Accrual Rates
Description: Percent of families approached who agreed to participate. This was done at the parent/dyad level.
Time Frame: 6 weeks after baseline
Population: This number refers to the parent-child dyads.
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 30 | 30
Participants | 24 | 24

3. Primary Outcome: Feasibility - Number of Participants Attending 75%+ Sessions
Description: Number of participants who completed at least 75% of the program sessions. This was done at the parent/dyad level.
Time Frame: 6 weeks after baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 47 | 48
Participants | 38 | 48

4. Primary Outcome: Retention Over Time (From Baseline to Post-assessment)
Description: Percentage of families retained for post-intervention assessment
Time Frame: From baseline to post-assessment (6-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 47 | 48
Participants | 44 | 35

5. Primary Outcome: Retention Over Time (From Baseline to 3-month Follow-up)
Description: Percentage of families retained for 3-month follow-up assessment
Time Frame: From baseline to 3-month follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 47 | 48
Participants | 41 | 35

6. Secondary Outcome: Child BMI z Score (Post-Assessment)
Description: Height (to the nearest 1/4 inch) using a metal ruler and weight (to the nearest 1/4 pound) using a scale will be measured by study staff.
  Z Body Mass Index (BMI). 0 represents the population mean. The higher the score, the higher the BMI, based on age and gender. There are no established clinically relevant thresholds for z-BMI.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 17
Z-score | 2.28 (.98) | 1.48 (1.02)

7. Secondary Outcome: Child BMI z Score (3-month Follow-up)
Description: as for outcome 6
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 19 | 16
Z-score | 2.30 (.83) | 1.58 (.89)

8. Secondary Outcome: Child Waist-to-Hip Ratio (Post-Assessment)
Description: Circumference of the hip (girth of hips above the gluteal fold) and waist (narrowest part of torso above the umbilicus and below the xiphoid process) will be measured by study staff using an anthropometric measuring tape and used to calculate continuous Waist-to-Hip Ratio.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: Waist-to-Hip Ratio
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 17
Waist-to-Hip Ratio | .92 (.05) | .92 (.07)

9. Secondary Outcome: Child Waist-to-Hip Ratio (3-month Follow-up)
Description: as for outcome 8
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: Waist-to-Hip Ratio
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 19 | 16
Waist-to-Hip Ratio | .94 (.09) | .90 (.08)

10. Secondary Outcome: Child Sugar Sweet Beverage and Fast Food Intake Instrument (Post-Assessment)
Description: The questionnaire consists of 11 questions on food and physical activity behaviors for youth participants in the study. This was adapted from the Youth Expanded Food and Nutrition Education Program (EFNEP) evaluation tool, the EFNEP 3rd-5th Grade Survey, which was designed and tested by Purdue University Extension Program. It will take approximately 5 minutes to complete. Below are presented the minimum and maximum values for each subscale reported.
  Fruit & Veg Frequency: 0-15, higher scores mean fruits and veggies consumed more frequently.
  Fruit & Veg Quantity: 0-5, higher scores mean larger fruit and veggie quantity consumed.
  Sugar-Sweetened Beverage Frequency: 0-8, higher scores mean SSB consumed more frequently.
  Sugar-Sweetened Beverage Quantity: 0-5, higher scores mean larger quantities of SSB consumed.
  Fast Food Frequency: 0-4, higher scores mean fast food consumed more frequently.
  Fast Food Quantity: 0-16, higher scores mean larger quantities of fast food consumed.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 17
score on a scale
  Fruit & Vegetable: Frequency | 7.18 (3.38) | 6.53 (2.35)
  Fruit & Vegetable: Quantity | 3.09 (.70) | 3.15 (.61)
  Sugar-Sweetened Beverage: Frequency | 2.23 (1.95) | 1.71 (1.36)
  Sugar-Sweetened Beverage: Quantity | 2.17 (1.30) | 1.91 (1.18)
  Fast Food: Frequency | .91 (.92) | .35 (.49)
  Fast Food: Quantity | 3.38 (2.96) | 1.53 (2.27)

11. Secondary Outcome: Child Sugar Sweet Beverage and Fast Food Intake Instrument (3-month Follow-up)
Description: The questionnaire consists of 11 questions on food and physical activity behaviors for youth participants in the study. This was adapted from the USDA Youth Expanded Food and Nutrition Education Program (EFNEP) evaluation tool, the EFNEP 3rd-5th Grade Survey, which was designed and tested by Purdue University Extension Program. It will take approximately 5 minutes to complete. Below are presented the minimum and maximum values for each subscale reported.
  Fruit & Veg Frequency: 0-15, higher scores mean fruits and veggies consumed more frequently.
  Fruit & Veg Quantity: 0-5, higher scores mean larger fruit and veggie quantity consumed.
  Sugar-Sweetened Beverage Frequency: 0-8, higher scores mean SSB consumed more frequently.
  Sugar-Sweetened Beverage Quantity: 0-5, higher scores mean larger quantities of SSB consumed.
  Fast Food Frequency: 0-4, higher scores mean fast food consumed more frequently.
  Fast Food Quantity: 0-16, higher scores mean larger quantities of fast food consumed.
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 19 | 16
score on a scale
  Fruit & Vegetable: Frequency | 5.84 (2.59) | 6.88 (3.01)
  Fruit & Vegetable: Quantity | 2.95 (.96) | 3.25 (.61)
  Sugar-Sweetened Beverage: Frequency | 1.63 (1.07) | 1.75 (1.34)
  Sugar-Sweetened Beverage: Quantity | 1.53 (.87) | 1.47 (1.01)
  Fast Food: Frequency | .74 (.56) | .75 (.86)
  Fast Food: Quantity | 3.26 (3.07) | 3.00 (2.63)

12. Secondary Outcome: Parent BMI (Post-Assessment)
Description: Height (to the nearest 1/4 inch) using a metal ruler and weight (to the nearest 1/4 pound) using a scale will be measured by the study staff and used to calculate continuous adult BMI score.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 18
kg/m^2 | 31.29 (4.59) | 30.86 (6.14)

13. Secondary Outcome: Parent BMI (3-month Follow-up)
Description: as for outcome 12
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 19
kg/m2 | 31.06 (4.47) | 31.41 (5.27)

14. Secondary Outcome: Parent Waist-to-Hip Ratio (Post-Assessment)
Description: Circumference of the hip (girth of hips above the gluteal fold) and waist (narrowest part of torso above the umbilicus and below the xiphoid process) will be measured by the study staff using an anthropometric measuring tape and used to calculate continuous Waist-to-Hip Ratio.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: Waist-to-Hip Ratio
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 18
Waist-to-Hip Ratio | .87 (.04) | .88 (.08)

15. Secondary Outcome: Parent Waist-to-Hip Ratio (3-month Follow-up)
Description: as for outcome 14
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: Waist-to-Hip Ratio
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 19
Waist-to-Hip Ratio | .88 (.08) | .88 (.07)

16. Secondary Outcome: Latino Dietary Behaviors Questionnaire (Post-Assessment)
Description: The Latino Dietary Behaviors Questionnaire: This 13-item self-report survey of dietary habits (in Spanish) assesses 4 areas of eating behavior -- healthy dietary changes; types of drinks consumed, number of meals per day and fat consumption. Minimum and maximum scores possible for this scale range from 1 to 47. Higher scores reflect healthier eating behaviors.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 18
score on a scale | 27.41 (4.58) | 26.00 (4.21)

17. Secondary Outcome: Latino Dietary Behaviors Questionnaire (3-month Follow-up)
Description: as for outcome 16
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 19
score on a scale | 26.59 (3.50) | 24.50 (3.43)

18. Secondary Outcome: Perceived Stress Scale (PSS) [Post-Assessment]
Description: Parents complete the 14 item self-report scale that asks participants about their feelings in the past month. Minimum and maximum scores possible for this scale range from 0 to 40. Higher scores reflect greater perceived stress.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 18
score on a scale | 16.27 (4.87) | 15.33 (4.91)

19. Secondary Outcome: Perceived Stress Scale (PSS) [3-month Follow-up]
Description: as for outcome 18
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 19
score on a scale | 15.36 (5.39) | 18.44 (2.50)

20. Secondary Outcome: Recognize Subscale of the Mindful Eating Questionnaire (Post-Assessment)
Description: Parents will complete the Recognize subscale of the Mindful Eating Questionnaire. The subscale has 9 items and is designed to assess an individual's ability to stop eating when full. Minimum and maximum scores possible for this subscale range from 9 to 36. Higher scores reflect a greater degree of recognition of hunger and satiety cues.
Time Frame: Post-Assessment (6 weeks after Baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 18
score on a scale | 30.55 (2.96) | 29.72 (2.74)

21. Secondary Outcome: Recognize Subscale of the Mindful Eating Questionnaire (3-month Follow-up)
Description: as for outcome 20
Time Frame: 3-month Follow-up (3 months after Post-Assessment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 22 | 19
score on a scale | 31.14 (4.72) | 29.13 (4.36)

ADVERSE EVENTS:
Time Frame: 19 weeks
Description: NIH's definition of adverse events.
Arm/Group | Feasibility and Acceptability of ADAPT+ | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/48
Other Adverse Events (participants affected / at risk) | 0/47 | 0/48

LIMITATIONS AND CAVEATS:
This study was a feasibility and acceptability pilot and was not powered to test the efficacy of our intervention, ADAPT+. The study results are preliminary in nature. Other key limitations are that participating parents primarily were mothers and that the study was geographically limited to only two rural communities where the project was implemented. COVID-19 also affected some of the recruitment efforts and did, at times, impact participant's attendance to sessions and assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04800432/Prot_SAP_000.pdf